CLINICAL TRIAL: NCT06081634
Title: Study on the Efficacy of a Psychological Approach for the Enhancement of Cognitive Reserve in a Bipolar Population With a Recent First Episode
Brief Title: Study Efficacy of Enhancing Cognitive Reserve in Patients With a First Bipolar Episode
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: FIDMAG Germanes Hospitalàries (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI18/00810
Record Dates: First submitted 2023-09-20; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Bipolar Disorder
Keywords: Cognitive reserve
MeSH Terms: conditions — Bipolar Disorder | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Experimental, multicentre, randomised, test-retest and control group clinical study to evaluate the efficacy of a cognitive reserve enhancement programme in patients with a diagnosis of bipolar disorder or schizoaffective disorder whose first episode has occurred within the last five years. Patients will be randomised into two groups: one group of patients will receive a psychological intervention for cognitive enhancement and another group of patients will receive only the usual pharmacological treatment (TAU).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhancing cognitive reserve (Active Comparator): After the baseline assessment, subjects will be randomly assigned by non-research staff, following the balanced clocks method, to receive a psychological intervention for the improvement of cognitive reserve (N=60) or to the group receiving TAU only (N=60). All assessments will be common to both groups. The experimental group will receive an intervention consisting of 12 weekly sessions of approximately 60 minutes duration. The aim of this intervention is to offer a series of strategies to increase academic and/or work achievements, leisure and free time activities, as well as an improvement in the level of neurocognitive functioning. Most of the tasks to be carried out are based on the use of pencil and paper with audiovisual support. Patients will also receive pharmacological follow-up in each center. A psychologist blind to the results of the assessment will provide the therapeutic approach for the improvement of cognitive reserve.
  Interventions: Behavioral: Enhancing cognitive reserve
- Placebo group (Placebo Comparator): This group will receive only pharmacological treatment supervised by the Psychiatrists of each Unit.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Enhancing cognitive reserve — Intervention in group format (6-8 patients) consisting of 12 weekly sessions, each lasting approximately 60 minutes. The aim of this intervention is to offer a series of strategies to increase academic and/or work achievements, leisure and free time activities, as well as an improvement in the level of neurocognitive functioning. Most of the tasks to be carried out are based on the use of pencil and paper with audiovisual support. Technological resources such as the use of the Internet and some telephone applications will also be used in some sessions. For those sessions in which the practice of mindfulness techniques will be promoted, a virtual reality device will be used per patient.
  Arms: Enhancing cognitive reserve
Other: Treatment as Usual — The group will only receive the pharmacoloical treatment according to the based guidelines.
  Arms: Placebo group

SUMMARY:
This study aims to adapt and apply a psychological program aimed at improving cognitive reserve (CR) in bipolar patients who have recently presented a first episode of the illness. The purpose of this project is to test both the effectiveness of the psychological intervention as well as the stability of the obtained results after nine months of follow-up. One-hundred and twenty patients (60 patients each centre) will be recruited and assessed with clinical, functioning, quality of life, neuropsychological and RC assessment tools. Then, participants will be randomly assigned to two different conditions: the experimental one, consisting in the implementation of the psychological intervention aiming at improving CR (n=60), and the control one, in which the usual pharmacological treatment will be carried on (n=60). Once the psychological intervention has finished (3 months) re-assessment of all the explored variables at baseline will be performed. Finally, after 12 months from the baseline visit, a re-assessment of all the participants in the study will be carried out to verify that post-intervention obtained results remain stable throughout the complete follow-up period. The investigators hypothesized that patients with a recent first episode who have undergone the intervention program will improve their CR as well as measures related to the severity of the difficulties observed at baseline concerning clinical, functioning, quality of life and neurocognitive performance. A second hypotheses is that all these changes will remain stable after nine month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 40 years of age whose disease onset (first episode) is within the last 5 years.
* Fulfill diagnostic criteria for bipolar disorder (type I or type II) or schizoaffective disorder, bipolar type, according to the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association (DSM-5) based on a semi-structured clinical interview.
* Patients in clinical remission or partial remission at the time of assessment, defined as scores ≤ 10 on the Young Mania Rating Scale (YMRS) (Young, 1978) and ≤ 14 points on the Hamilton Depression Rating Scale (HAMD) (Hamilton, 1960).
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Estimated IQ less than 85.
* Any medical condition that may affect neuropsychological performance (such as neurological diseases).
* Presence of any comorbid psychiatric condition (except substance use/abuse).
* Patients who have received any type of psychological intervention in the 6 months prior to the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Cognitive reserve | one year
  Assess cognitive reserve, a potential mechanism to cope with brain damage. Assessed by the Cognitive Reseve Assessment Scale (CRASH), (Amoretti et al, 2019). The CRASH scale provides a global score and a score for each of the domains that form it (education, occupation, and intellectual and leisure activities). The scale's maximum total score is 90, and it can be calculated using a formula, created with the intention that all domains have the same weighting in the final score. The score for each domain is obtained by adding the scores of the items it contains. For all scores, the higher the result, the better the level of cognitive reserve. .

SECONDARY OUTCOMES:
Depressive symptoms | one year
  Assess the clinical state (depressive symptoms) of the patients pre and post intervention.
  The depressive symptoms will be assessed by the Hamilton Depression Rating Scale (HDRS). For the 17-item version, a score of 0-7 is considered to be normal while a score of 20 or higher (indicating at least moderate severity). The total score ranges from 0 to 52. Each question has between three and five possible answers, with a score of 0-2 or 0-4 respectively.
  The manic symptoms will be assessed by the Young Mania Rating Scale (YMRS) (Young, 1978) which is a gold-standard clinician-rated assessment tool for severity of manic symptoms. The total YMRS scores ranges from 0 to 60, with higher scores indicating more severe mania.
Manic symptoms | one year
  Assess the severity of manic symptoms of the patients pre and post intervention.
  The manic symptoms will be assessed by the Young Mania Rating Scale (YMRS) (Young, 1978) which is a gold-standard clinician-rated assessment tool for severity of manic symptoms. The total YMRS scores ranges from 0 to 60, with higher scores indicating more severe mania.
Number of participants with subjective cognitive complaints | One year
  Related cognitive concerns expressed by people with or without objective evidence of cognitive impairment. It will be assessed by the Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA) The COBRA utilizes queries informed by everyday mental tasks. Sixteen items, including verbal learning and memory, executive functionality, attention/concentration, working memory, processing speed, and mental tracking, are used to measure subjective cognitive dysfunction,14 and a four-point scale is used to rate these items (0 = never, 1 = sometimes, '2 = often, and 3 = always). The total COBRA score is calculated by adding the rating of each item; the highest possible score is 48, and scores of ≥15 indicate moderate to severe subjective cognitive impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain